CLINICAL TRIAL: NCT03515655
Title: Characterizing Acute Heart Failure With Reduced Ejection Fraction Hospitalization Outcomes
Brief Title: A Study of Patients Hospitalized With Acute Heart Failure With Reduced Ejection Fraction (HFrEF)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV013-029
Record Dates: First submitted 2018-04-23; First posted 2018-05-03 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A study of participants hospitalized with acute heart failure with reduced ejection fraction

ELIGIBILITY:
Inclusion Criteria:

* An average left ventricular ejection fraction (LVEF) < 40% over the entire index hospitalization
* Age 18 years or older on the index date
* At least 6 months of activity in the databaseprior to the index date

Exclusion Criteria:

* Any code for myocardial infarction (ICD-9 diagnosis code: 410.xx, ICD-10 diagnosis code: I21.xx) or related terms such as "myocardial infarction", "mi", "infarct" or "heart attack" occurring during the index hospitalization

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be patients who were hospitalized with acute heart failure with an average reduced ejection fraction≤40during hospitalization, and who do not have a coincident myocardial infarction and who have at least 6 months of activity in the database prior to the hospitalization.
Sampling Method: Probability Sample
Enrollment: 99209 (Estimated)
Dates: Start 2018-02-21 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of 30 day mortality | 30 days
Incidence of 30 day readmission | 30 days
Incidence of a prolonged length of stay | 30 days
Incidence of participants hospitalized with AHF with reduced ejection fraction | 6 years

SECONDARY OUTCOMES:
Distribution of socio-demographic characteristics in participants hospitalized for acute HFrEF | 6 years
  Socio-demographic characteristics will be summarized using descriptive statistics
Distribution of clinical characteristics in participants hospitalized for acute HFrEF | 6 years
  Clinical characteristics will be summarized using descriptive statistics

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Princeton, New Jersey, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx